CLINICAL TRIAL: NCT01420562
Title: Pharmacokinetics of Posaconazole in Allogeneic Transplant Patients With Mucositis
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML7267
Record Dates: First submitted 2011-08-16; First posted 2011-08-19 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: allogeneic HSCT; posaconazole; prophylaxis; mucositis; pharmacokinetics
MeSH Terms: conditions — Mucositis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Posaconazole oral suspension: One group of patients will receive posaconazole oral suspension as prophylactic agent.
  Blood sampling: At day of transplantation, day 7 and 14, 9 blood samples will be collected to calculate AUC. Moreover, citrulline will be determined to objectively evaluate the severity of mucositis.
  Interventions: Procedure: blood sampling
- Posaconazole oral tablet: Once the oral tablet is available for adminstration to patients, a second group of patients will receive these tablets as prophylactic agent.
  Blood sampling: At day of transplantation, day 7 and 14, 9 blood samples will be collected to calculate AUC. Moreover, citrulline will be determined to objectively evaluate the severity of mucositis.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — During posaconazole treatment, blood sampling will occur on day 0 (=day of transplantation), day 7 and 14 to correlate posaconazole exposure to severity of mucositis.

SUMMARY:
The goal of this study is to calculate pharmacokinetic parameters and to evaluate the trough levels of posaconazole reached in patients with different stages of mucositis, due to chemotherapy and total body irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving allogeneic stem cell transplantation - Treated with prophylactic posaconazole: oral suspension (200mg three times daily) or tablet (300mg once daily) to prevent invasive fungal infections

Exclusion Criteria:

* Gastroparesis
* Vomiting or diarrhea within 2 hours after intake of posaconazole
* Concomitant administration of potent inducers of the enzyme UGT1A4: carbamazepine,phenytoin, phenobarbital, rifabutin, rifampicin,...
* Age under 18 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the hematology ward who will receive an allogeneic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2011-09; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Posaconazole plasma levels and area under the curve in patients with different stages of mucositis | Day 0 (day of transplantation), day +7, day +14
  Plasma levels of posaconazole will be determined to calculate the area under the curve. These values will be correlated with the stage of mucositis, which will be assessed using citrulline monitoring in plasma. The stage of mucositis will also be assessed using the Daily Oral Mucositis Score (DMS) and Daily Gut Mucositis Score (DGS).

CONTACTS AND LOCATIONS:
Overall Officials: Kim Vanstraelen, R.Ph., Principal Investigator — Catholic University of Leuven, Faculty of Pharmacy, division Hospital Pharmacy
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium